CLINICAL TRIAL: NCT03038243
Title: A Phase 2a/2b, Randomized, Double-blinded, Placebo-controlled, Trial to Assess the Safety, Immunogenicity and Efficacy of Inactivated Shigella Flexneri 2a Whole Cell (Sf2aWC) Vaccine Administered With and Without Double Mutant E. Coli Heat Labile Toxin (dmLT) in Healthy Adult Subjects
Brief Title: Safety, Immunogenicity and Efficacy Study of Inactivated Whole Cell Shigella Flexneri 2a Vaccine With and Without dmLT in Adults
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: PATH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VAC-047
Record Dates: First submitted 2017-01-23; First posted 2017-01-31 (Estimated); Last update posted 2017-11-20 (Actual); Status verified 2017-11

CONDITIONS: Shigella Sonnei Dysenteries
Keywords: Shigella; vaccine; shigellosis; dysentery; whole cell
MeSH Terms: conditions — Dysentery, Bacillary; Dysentery | interventions — Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Experimental): Group 1, 2.25 x 10^11 Sf2aWC cells +10 µg dmLT Group 2, 2.25 x 10^11 Sf2WC cells Group 3, 2.0 grams of NaHCO3 dissolved in 150 mL of sterile water
  Interventions: Biological: Shigella flexneri 2a whole cell (Sf2aWC) vaccine and double mutant E. coli heat labile toxin (dmLT); Biological: Shigella flexneri 2a whole cell (Sf2aWC) vaccine; Other: Placebo
- Cohort 2 (Experimental): Group 1, 2.25 x 10^11 Sf2aWC cells +10 µg dmLT Group 2, 2.25 x 10^11 Sf2WC cells Group 3, 2.0 grams of NaHCO3 dissolved in 150 mL of sterile water
  Interventions: Biological: Shigella flexneri 2a whole cell (Sf2aWC) vaccine and double mutant E. coli heat labile toxin (dmLT); Biological: Shigella flexneri 2a whole cell (Sf2aWC) vaccine; Other: Placebo
- Cohort 3 (Experimental): Group 1, 2.25 x 10^11 Sf2aWC cells +10 µg dmLT Group 2, 2.25 x 10^11 Sf2WC cells Group 3, 2.0 grams of NaHCO3 dissolved in 150 mL of sterile water
  Interventions: Biological: Shigella flexneri 2a whole cell (Sf2aWC) vaccine and double mutant E. coli heat labile toxin (dmLT); Biological: Shigella flexneri 2a whole cell (Sf2aWC) vaccine; Other: Placebo

INTERVENTIONS:
Biological: Shigella flexneri 2a whole cell (Sf2aWC) vaccine and double mutant E. coli heat labile toxin (dmLT) — 2.25 x 10^11 Sf2aWC cells +10 µg dmLT administered orally on Days 0, 28, and 56
Biological: Shigella flexneri 2a whole cell (Sf2aWC) vaccine — 2.25 x 10^11 Sf2WC cells administered orally on Days 0, 28, and 56
Other: Placebo — 2.0 grams of NaHCO3 dissolved in 150 mL of sterile water

SUMMARY:
This is a research study about an experimental (investigational) oral inactivated whole cell Shigella flexneri 2a killed vaccine (Sf2aWC) and an adjuvant called dmLT. Sf2aWC is a killed vaccine that is being made to prevent disease from Shigella., which causes bloody, watery diarrhea. An adjuvant is something that is added to a vaccine to make it work better. The purpose of the study is to see if the vaccine will protect people from Shigella infection with or without an adjuvant called dmLT. About 72 healthy adults, ages 18-45, will participate in this study. The study will compare 2 different vaccination groups and 1 control group. Volunteers have an equal chance to be in any of the 3 groups. Study procedures include: stool samples, blood samples and documenting side effects. Participants will be involved in study related procedures for about 6 months.

DETAILED DESCRIPTION:
Despite the public health burden of Shigella spp. on travelers, deployed soldiers and, most significantly, young children in the developing world, there is no licensed vaccine against Shigella. The rationale for using Shigella flexneri 2a whole cell killed vaccine (Sf2aWC), is that it is expected to be especially well tolerated by subjects. This is a single site, 2a/2b, double-blind, randomized, placebo-controlled, study in healthy adult subjects. Approximately 72 subjects will be enrolled into one of three vaccination groups: Sf2aWC 1011 Sf2aWC cells plus 10 µg dmLT (Group 1, n=24), 1011 Sf2WC cells alone (Group 2, n=24); or placebo (Group 4, n=24). The placebo preparation will be bicarbonate buffer.

After the vaccination phase subjects will be admitted by cohort on day 84 to an inpatient facility for 12 days to undergo challenge with approximately 1500 colony forming units (CFU) of wild type S. flexneri 2a strain 2457T (administered with NaHCO3 buffer). After 5 days of observation for clinical endpoints (or earlier and within 12 hours if they meet the definition of moderate-to-severe shigellosis as defined in the primary endpoints section below), subjects will receive a 5-day course of orally administered ciprofloxacin.

The primary objective of this study are to 1) evaluate, the safety and reactogenicity of 3 oral sequential doses of Sf2aWC with or without dmLT, 2) To measure the protective efficacy of 3 spaced doses of high-dose Sf2aWC vaccine with and without dmLT against moderate-to-severe shigellosis following experimental oral challenge with wild-type S. flexneri 2a 2457T

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults, male or female, age 18 to 45 years (inclusive) at the time of enrollment.
2. General good health, without clinically significant medical history, physical examination findings or clinical laboratory abnormalities per clinical judgment of PI.
3. Willingness to participate in the study after all aspects of the protocol have been explained and written informed consent obtained.
4. Completion of a training session and demonstrated comprehension of the protocol procedures and knowledge of Shigella associated illness by passing a written examination (70% pass score).
5. Availability for the study duration, including all planned follow-up visits.

Exclusion Criteria:

1. Presence of a significant medical or psychiatric condition that in the opinion of the investigator precludes participation in the study. Some medical conditions that are adequately treated and stable would not preclude entry into the study. These conditions might include stable asthma controlled with inhalers or mild hypertension stably controlled with a single agent.
2. Significant abnormalities in screening hematology, or serum chemistry as determined by PI or PI in consultation with the Medical Officer and sponsor.
3. Recent of a non-study vaccine or receipt of another investigational product (within 14 days before vaccination).
4. Have household contacts who are <3 years old or >70 years old or infirm or immunocompromised (for reasons including corticosteroid therapy, HIV infection, cancer chemotherapy, or other chronic debilitating disease).
5. Use of any medication that affects the immune function (e.g., corticosteroids and others) within 30 days preceding the first vaccination or planned use during the active study period.
6. Symptoms of Traveler's diarrhea associated with travel to countries where Shigella or other enteric infections are endemic (most of the developing world) within 1 year prior to dosing.
7. History of shigellosis or Shigella vaccination or challenge or a laboratory worker with known exposure to Shigella within the last 6 months
8. Prior receipt of experimental Shigella vaccine or live Shigella challenge within 3 years.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2017-08-01 (Estimated); Primary Completion 2018-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
solicited reactions, AEs, SAEs | first vaccination through 6 months post-3rd vaccination
  solicited reactions, AEs, SAEs assessed post-vaccination using targeted physical examinations, vital signs, and clinical laboratory tests
prevention of moderate to severe shigellosis | up to 24 hours
  prevention of moderate to severe shigellosis identified by diarrhea, fever, dysentery, and other signs/symptoms of enteric illness

CONTACTS AND LOCATIONS:
Overall Officials: Wilbur Chen, MD, MS, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- Center for Vaccine Development (CVD), University of Maryland School of Medicine, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No